CLINICAL TRIAL: NCT03163771
Title: Evaluation of a New Strategy for the Diagnosis of Peroxisomal Diseases
Acronym: PEROXY4G
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2015_12; 2016-A01147-44 (Other: ID-RCB number, ANSM); PHRCI_2014 (Other: PHRC number, DGOS)
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Peroxisomal Disorders; Diagnoses Disease
MeSH Terms: conditions — Peroxisomal Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The principal aim of the study is to avoid the diagnostic wanderings of patients suffering from a peroxisomal disorder. For this purpose, a new diagnostic strategy is proposed. It rests on functional metabolic explorations and gene studies directly connected to a first-line enlarged physico-chemical detection of metabolites from peroxisomal origin in clinically suspect patients.

ELIGIBILITY:
Inclusion Criteria:

I - CLINICAL/BIOLOGICAL CRITERIA For an efficient screening of the patients of the 4 contributing University Hospitals (Amiens, Caen, Lille and Rouen), various inclusion criteria were selected: In general, the inclusion criterion is the existence of a positive biology or in turn the persistence of a clinical suspicion in spite of a negative biology.

I A - Children from 0 to 17 years:

The clinical inclusion criterion is a positive biology or the persistence of a clinical suspicion in spite of a negative biology. This persistent clinical suspicion is left to the discretion of the clinician. It is essentially based on the existence of a family history of peroxisomal (or suspected) pathology and / or the combination of several clinical signs of craniofacial dysmorphism, skeletal abnormalities, encephalopathy (seizures, ataxia, Hypotonia), demyelinating peripheral neuropathy, ophthalmopathy (retinopathy, cataract), hepatic impairment (hyperbilirubinemia, hepatomegaly, cholestasis) and growth retardation OR I B - Adults from 18 years

The neurological symptoms of peroxisomal diseases in adulthood are numerous and non-specific. The three inclusion criteria selected for patient selection are as follows:

* Cognitive impairment (delayed acquisition or regression) and / or leukodystrophy AND At least one of the following signs: Cerebellar ataxia, Spastic paraparesis, Peripheral neuropathy, Neurosensory deafness, Retinitis pigmentosa, Epilepsy, Unexplained unexplained vigilance, Peripheral corticotropic insufficiency +/- gonadotropic AND
* no evidence for an extraperoxisomal origin of the patient disease stated after the usual paraclinic explorations

II - NON CLINICAL CRITERIA

* Social insurances
* Having understood the information note and having signed the informed consent form.
* Patients under guardianship or curatorship may be included, since peroxisomal diseases as a cause of neurological impairment may potentially lead to guardianship.

Exclusion Criteria:

* Pregnant or nursing women
* Person deprived of liberty or in emergency situations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The studied population is represented by only one group of patients checking the inclusion criteria and recruited in the 4 University Hospital centers (Amiens, Caen, Lille and Rouen). For each patient, diagnostic exploration will start in patients with the common inclusion criteria and will include the study of all biochemical parameters susceptible to be disturbed In peroxisomal pathologies (Biology component). Based on the data obtained, the inclusion of patients will lead to biological confirmation tests (Cell Exploration and Enzymology) and molecular studies (Molecular Biology).
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Percentage of cases diagnosed by the new procedure versus the number of patients included. | 14 months
  Evaluation of a diagnostic strategy based on functional metabolic explorations and gene studies directly connected to a first-line enlarged physico-chemical detection of metabolites from peroxisomal origin in clinically or biologically suspect patients
  The study is concomitant with an implementation in the routine Hospitals of the inter-region (West and North of France) of an immediate wide exploration (and not sequential and optional) of diagnostic markers of a pathology peroxisomal. This wide exploration should by itself lead to a diagnosis enrichment and should increase the number of inclusions. But the study, for patients thus included, is also considering an enlarged scanning of functional and genetic explorations that follow inclusion (instead of targeted screening guided primarily by the biological anomaly in the usual practice).

SECONDARY OUTCOMES:
Number of new cases diagnosed by the new procedure in relation to the number of habitants per year. | 14 months
  Evaluation of a diagnostic strategy based on functional metabolic explorations

CONTACTS AND LOCATIONS:
Overall Officials: Joseph VAMECQ, MD, Principal Investigator — University Hospital, Lille
Locations (4):
- France (4):
  - Département de Pédiatrie, Unité de Génétique Clinique, CHU d'Amiens, Amiens
  - Pédiatrie, CHU Clémenceau de Caen, Caen
  - Hôpital Jeanne de Flandres, CHRU, Lille
  - Pédiatrie, Pavillon Mère et Enfant, CHU Ch. Nicolle de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No